CLINICAL TRIAL: NCT00844766
Title: A Study to Validate a Home-screening Test for Lactose Intolerant People
Brief Title: Validation of a Home-screening Test for Lactose Intolerance
Status: Withdrawn | Type: Observational
Why Stopped: This study was stopped as no patient asked to participate was prepared to do so
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Carolyn Burden, University Hospitals of Leicester NHS Trust
Other Study IDs: UHL 10268
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Lactose Intolerance
Keywords: Lactose intolerance; Lactose; Home-screening test; Validate
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The hypothesis underlying this study is that whilst there is no home-screening test for lactose intolerance, this test would have significant value as lactose tolerance tests and breath hydrogen tests are expensive and time consuming. Therefore, it would be highly beneficial to validate a simple home-screening test.

This study will validate a simple home-screening test that uses lactose and not milk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed lactose intolerance as demonstrated by a lactose tolerance test
* Diagnosed as not having lactose intolerance as demonstrated by a lactose tolerance test

Exclusion Criteria:

* Pregnant
* Breastfeeding
* Unwillingness to comply with study outline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with lactose intolerance
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Mayberry, DSc MD, Principal Investigator — University Hospitals, Leicester